CLINICAL TRIAL: NCT06415929
Title: Single-center Retrospective Study Evaluating the Characteristics, Quality of Life and Satisfaction of Patients Undergoing Nail Resection With Dermal Matrix and Skin Graft Reconstruction at Nice University Hospital.
Brief Title: Etude rétrospective Monocentrique MATRIX
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 24Chirplast04
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-03

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with history: Patient with history of complete exeresis of the nail apparatus, with dermal matrix repair and total skin grafting

SUMMARY:
"Monocentric retrospective study.Analysis of a case series of patients who underwent nail resection with dermal matrix and skin graft reconstruction in the setting of nail bed malignancy.

Objective: To assess patients' quality of life and satisfaction with the function and aesthetics of dermal matrix and skin graft reconstruction of the nail apparatus.

Monocentric retrospective study.Analysis of a case series of patients who underwent nail resection with dermal matrix and skin graft reconstruction in the setting of nail bed malignancy.

Objective: To assess patients' quality of life and satisfaction with the function and aesthetics of dermal matrix and skin graft reconstruction of the nail apparatus.

"

ELIGIBILITY:
Inclusion Criteria:

- Adult patients who have undergone complete nail removal for malignancy - Reconstructed with INTEGRA dermal matrix and total skin graft.

Exclusion Criteria:

-Minor patients -Patients who have undergone complete removal of the nail apparatus for malignancy but have been reconstructed in another way (flap, isolated skin graft)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hopital de soins tertiaires- Hopital Pasteur 2-Nice
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Quality of life evaluation | 3 months too 36 months after the surgery
  Quality of life evaluation- questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Elise Elise, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU NiICE, Nice, Alpes Maritimes, France